CLINICAL TRIAL: NCT06897865
Title: The Effect of Pressure Sore Preventıon Traınıng Wıth Vırtual Realıty on Satisfaction and Self-Confıdence Perceptıon in Nursıng Students
Brief Title: Nursing Students Education Virtual Reality Wound Care
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Murat Çağatay Sonkaya, LECTURER, Ankara Medipol University
Other Study IDs: 07/864
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Nurse's Role; Wound Heal; Prevention
Keywords: nursing; virtual reality; wound care
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: 35 students in the experimental group will first be administered the "Knowledge Assessment Form for Pressure Sore Prevention" together with all participants. Then, these students will be given pressure sore training using virtual reality (VR) goggles. After the training, the same assessment form will be applied again to measure their learning level. Students' perceptions of the training process will be assessed with the "Student Satisfaction and Self-confidence in Learning Scale". Finally, the "Knowledge Assessment Form for Pressure Ulcer Prevention" will be administered to the students again after three months to determine the long-term effect of the training.
  Interventions: Other: survey
- control group: In the first stage, 35 students in the control group will be administered the "Knowledge Assessment Form for Pressure Sore Prevention" together with all participants. Then, an informative booklet about pressure sores will be given to the students in this group. After the training provided with the booklet, the same assessment form will be applied again to measure their level of knowledge. The satisfaction and self-confidence levels of the students regarding the education process will be evaluated with the "Student Satisfaction and Self-Confidence in Learning Scale". In the final stage, the "Knowledge Assessment Form for Pressure Ulcer Prevention" will be applied again after three months to measure the retention of knowledge.
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — SURVEY

SUMMARY:
This study is a randomized controlled trial aiming to determine the effect of pressure sore prevention education given to nursing students at a foundation university through virtual reality on student satisfaction, self-confidence perception and knowledge retention. The study will investigate whether virtual reality training affects student satisfaction and self-directed learning skills, differences between pre-test and post-test scores, and retention of the training. 66 nursing students will be included in the study, the experimental group will be trained with VR goggles and the control group will be provided with written material. The data obtained during the data collection process will be analyzed with the SPSS V23.0 program, descriptive statistics and appropriate parametric or nonparametric tests will be used. The measurement tools to be used include the 20-question "Knowledge Assessment Form for Pressure Ulcer Prevention" developed by Jeffries & Rizzolo and the "Student Satisfaction and Self-Confidence in Learning Scale". Ethics committee approval, relevant permissions and participant consent will be obtained for the study and the data obtained will be stored for 5 years and then destroyed. The literature review reveals the widespread use of virtual reality in education, healthcare and other fields and the critical role of pressure sore prevention in reducing healthcare costs and improving the quality of patient care.

DETAILED DESCRIPTION:
This study will be conducted as a pre-test post-test randomized controlled trial to determine the effect of pressure sore prevention education on student satisfaction, self-confidence perception, and knowledge retention at Ankara Medipol University Department of Nursing. Data will be collected from 70 nursing students through an online survey, the experimental group will be trained with VR goggles, while the control group will be provided with written material. Data collection will take place in five phases: pre-test, training, post-test, satisfaction and confidence assessment, and a retention test after three months. The measurement tools to be used include the 20-question "Knowledge Assessment Form for Pressure Ulcer Prevention" developed by Jeffries & Rizzolo and the "Student Satisfaction and Confidence in Learning Scale". Data will be analyzed in SPSS V23.0 and appropriate parametric or nonparametric tests will be applied. Data will be collected between March 2025 and July 2025 and will be stored for five years and then destroyed.

ELIGIBILITY:
İnclusion Criteria

* Nursing Students,
* 2nd year nursing student

Exclusion Criteria

* not a nursing student
* 1st, 3rd or 4th year nursing student

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: 70 nursing student
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-21 (Estimated); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Data collection | 1 week
  All students will be administered the "Knowledge Assessment Form for Pressure Ulcer Prevention".
VR application | 1 week
  35 students will be trained on pressure sores using virtual reality (VR) goggles.

IPD SHARING:
Plan to Share IPD: No